CLINICAL TRIAL: NCT00003137
Title: A Phase II Trial of CPT-11 in Patients With Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction Incorporating Pretreatment and Posttreatment Biopsies for Evaluation of Tumor Thymidylate Synthase, MIB-1, Topoisomerase I, and p53
Brief Title: Irinotecan in Treating Patients With Advanced Cancer of the Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-964152; CDR0000065905 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-01-22 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; stage IV esophageal cancer; adenocarcinoma of the esophagus; intestinal adenocarcinoma of the stomach; diffuse adenocarcinoma of the stomach; mixed adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan (Experimental): Patients receive irinotecan (CPT-11) by IV over 90 minutes every 3 weeks. Dosage modifications are made based on toxicity. Retreatment may be delayed another 3 weeks (for a total of 6 weeks) to allow for recovery from toxic effects. Patient is taken off study if they do not recover from toxic effects, unless cause is documented to be unrelated to CPT-11. Patients with stable disease or partial response continue on treatment until disease progression or intolerable toxicity. Patients with complete response continue on treatment for another 2 courses and then are observed.
  Patients are followed every 3 months for 3 years or until disease progression.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have advanced cancer of the stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate, survival, and toxicity of previously untreated patients with locally advanced or metastatic gastric cancer who are treated with irinotecan (CPT-11).

OUTLINE: This is a nonrandomized study. Patients receive irinotecan (CPT-11) by IV over 90 minutes every 3 weeks. Dosage modifications are made based on toxicity. Retreatment may be delayed another 3 weeks (for a total of 6 weeks) to allow for recovery from toxic effects. Patient is taken off study if they do not recover from toxic effects, unless cause is documented to be unrelated to CPT-11. Patients with stable disease or partial response continue on treatment until disease progression or intolerable toxicity. Patients with complete response continue on treatment for another 2 courses and then are observed. Patients are followed every 3 months for 3 years or until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced adenocarcinoma of the stomach or gastroesophageal junction beyond hope of surgical cure and not considered a candidate for potentially curative chemotherapy/radiation therapy Measurable or evaluable disease Tumor must be accessible for biopsy No known central nervous system metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 150,000/mm3 Hemoglobin at least 9.0 mg/dL (transfusion allowed) Hepatic: Bilirubin no greater than upper limit of normal (ULN), regardless of liver involvement secondary to tumor AST no greater than 3 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No unstable angina No uncontrolled high blood pressure No active congestive heart failure No myocardial infarction in the last 6 months No serious uncontrolled cardiac arrhythmia No New York Heart Association Class III or IV heart disease Pulmonary: No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung No pleural effusion or ascites, which cause respiratory compromise (at least Grade 2 dyspnea) Other: No active or uncontrolled infection No prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancer from which the patient has been disease free for at least 5 years Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for gastric or gastroesophageal junction cancer No prior irinotecan (CPT-11) or other camptothecin Endocrine therapy: Not specified Radiotherapy: No prior abdominal or pelvic radiotherapy No prior radiotherapy to greater than 25% of bone marrow No prior radiotherapy to measurable or evaluable indicator lesions At least 4 weeks since major radiotherapy (chest radiotherapy) Surgery: At least 3 weeks since major surgery and recovered At least 2 weeks since minor surgery and recovered Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 1997-12; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 3 years

SECONDARY OUTCOMES:
survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Goldberg, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Jatoi A, Foster NR, Egner JR, Burch PA, Stella PJ, Rubin J, Dakhil SR, Sargent DJ, Murphy BR, Alberts SR. Older versus younger patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and stomach: a pooled analysis of eight consecutive North Central Cancer Treatment Group (NCCTG) trials. Int J Oncol. 2010 Mar;36(3):601-6. doi: 10.3892/ijo_00000535. PMID 20126980
- [Result] Erlichman C, Goldberg RM, Mahoney MR, et al.: A phase II trial of CPT-11 in patients (pts) with advanced gastric or gastroesophageal (GE) junction adenocarcinoma (ADCA): a clinical and pharmacodynamic evaluation. A North Central Cancer Treatment Group (NCCTG) study. [Abstract] J Clin Oncol 23 (Suppl 16): A-4026, 314s, 2005.